CLINICAL TRIAL: NCT07266545
Title: RNA Editing as a Biomarker of Antidepressant Response in Unipolar and Bipolar Depression (EDIT-ANDRE)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aysegul Ozerdem, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-006875
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Unipolar Depression; Bipolar Depression
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder | interventions — Vortioxetine; cariprazine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vortioxetine (Experimental): Subjects randomized to the vortioxetine arm will begin 8 weeks of treatment with vortioxetine at 10 mg/day, titrated to 20 mg/day (after 7 days).
  Subjects who do not meet remission criteria will enter a second 8 week augmentation phase.
  Interventions: Drug: Vortioxetine; Drug: Cariprazine (Augmentation Phase)
- Bupropion (Experimental): Subjects randomized to the bupropion arm will begin 8 weeks of treatment with buproprion extended release at 150 mg/day; titrated to 300 mg/day (after 7 days)
  Subjects who do not meet remission criteria will enter a second 8 week augmentation phase.
  Interventions: Drug: Bupropion extended release; Drug: Cariprazine (Augmentation Phase)

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine, once daily, for 8 weeks
  Arms: Vortioxetine
Drug: Bupropion extended release — Bupropion extended release, once daily, for 8 weeks
  Arms: Bupropion
Drug: Cariprazine (Augmentation Phase) — Participants who do not meet remission criteria will enter a second 8-week augmentation phase (Weeks 9-16).
  During this phase, cariprazine will be added to the existing regimen, administered orally once daily in the morning, starting at 1.5 mg/day and titrated up to 3.0 mg/day in one week.

SUMMARY:
The purpose of this research is to understand how changes in RNA editing relate to treatment response in unipolar and bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Adult females and males, aged 18-65 years
* Must have the capacity to understand study procedures, to comply with them for the entire length of the study, and to provide informed consent.
* Current major depressive episodes associated with MDD, BD-I, or BD-II, confirmed using the SCID-IV-CV.
* Symptom severity score on the Quick Inventory for Depressive Symptomatology - Clinician (QIDS-C16) > 10.
* Ability to travel for assessment visits.
* Negative urine pregnancy test for people of childbearing potential
* People of childbearing potential must be using an acceptable method of birth control during the study, such as hormonal contraception, intrauterine device, bilateral tubal ligation, partner's documented vasectomy, or complete abstinence from intercourse with childbearing potential, with barrier methods permitted only when used in combination with one of these primary methods.
* BD-I patients must be on a mood stabilizer (i.e., lithium, valproate, or a mood-stabilizing atypical antipsychotic at least for one month) at the time of enrollment Exclusion Criteria

All candidates meeting any of the following criteria at baseline will be excluded from study participation:

* Individuals who cannot understand English will not be enrolled because informed consent, study procedures, and interviews require comprehension of English.
* Inability to provide written, voluntary informed consent
* Failure to score at least 75% on a 4-item comprehension assessment related to study goals, risks, and benefits
* For BD-I: not having used at least one mood stabilizer (e.g., lithium, valproate, or mood-stabilizing antipsychotics) at a stable dose and within a therapeutically effective antimanic range for a minimum of one month.
* History of treatment-refractory depression, defined as non-response to two or more antidepressant or mood-stabilizing regimens despite adequate dose, duration, and adherence during the current episode.
* Participants with active suicidal ideation, defined as a MADRS item #10 score greater than 4 or a "yes" response to item #4 (ideation with intent) or item #5 (ideation with plan) on the C-SSRS, will be excluded
* A medically serious suicide attempt within the past 6 months, defined as requiring emergency department evaluation, a medical procedure, or admission to a hospital (e.g., internal medicine, cardiology, or ICU)
* Current use of monoamine oxidase inhibitors or use within 14 days following discontinuation of a monoamine oxidase inhibitor
* Presence of mixed symptoms of depression, defined as a YMRS score ≥12
* Current use of any of the study medications (e.g., vortioxetine, bupropion, or cariprazine) at the time of enrollment (previous use of these medications is acceptable)
* Prior hypersensitivity reaction or documented non-response to any of the study medications
* A history of seizure disorder; complicated febrile convulsions (e.g., prolonged, focal, or recurrent); current or past diagnosis of bulimia nervosa or anorexia nervosa; or any condition known to lower seizure threshold, including abrupt discontinuation of alcohol, benzodiazepines, barbiturates, or antiepileptic drugs.
* Known CYP2D6 or CYP2B6 poor metabolizer status, or a history of intolerance to medications primarily metabolized by these enzymes (e.g., vortioxetine, bupropion, SSRIs, efavirenz), due to increased risk of side effects.
* Recent use (within the past 4 weeks) of long half-life psychotropic medications with active metabolites that may interfere with study outcomes, including fluoxetine and long-acting injectable forms of aripiprazole and paliperidone.
* Active psychosis, defined as a YMRS item #8 score >4 or diagnosis of schizophrenia, schizoaffective disorder, delusional disorder, or schizophreniform disorder as determined by structured clinical interview
* Current drug or alcohol use disorder (excluding nicotine); full remission for at least 3 months is required for eligibility
* Positive toxicology screen for illicit substances (e.g., cocaine, methamphetamine, illegal opiates). Participants who use cannabis for recreational or medicinal purposes and fail the toxicology screen can potentially be included in the study only if they take the CUDIT-R and score a 12 or less.
* Individuals who are pregnant, lactating, trying to conceive, or not using adequate contraception (e.g., hormonal contraception, intrauterine device, tubal ligation, or condoms)
* Any active or unstable medical condition judged by the principal investigator to confer excessive risk
* Clinically significant laboratory abnormality, uncontrolled hypertension (blood pressure >160/100 mmHg), or tachycardia (heart rate >110 bpm)
* Significant renal, hepatic, or cardiac disease; malignancy; autoimmune disease; or chronic kidney disease > stage IIIa (estimated GFR < 60 mL/min/1.73 m²)
* History of traumatic brain injury or gastric bypass
* Clinical diagnosis of delirium, encephalopathy, intellectual disability or cognitive disorder (mild or major neurocognitive disorder)
* Currently receiving electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), vagus nerve stimulation (VNS), or deep brain stimulation (DBS) as acute or maintenance treatment
* Current use of systemic steroids, chemotherapy, radiotherapy, or undergoing involuntary psychiatric hospitalization
* Daily use of lorazepam (Ativan) >4 mg/day, or equivalent doses of other benzodiazepines (e.g., clonazepam >1 mg, alprazolam >2 mg, diazepam >20 mg)
* No access to smartphones, internet

All candidates meeting any of the following criteria at baseline will be excluded from the Phase 2 (cariprazine add-on) of the study:

* Meeting symptomatic remission criteria based on MADRS (≤ 10).
* Current use of a strong or moderate CYP3A4 inhibitor (e.g., ketoconazole, clarithromycin, fluconazole, or verapamil) or a strong CYP3A4 inducer (e.g., carbamazepine, rifampin, phenytoin, or St. John's Wort), due to potential pharmacokinetic interactions with cariprazine.
* Diagnosis of BD-I with concurrent use of an antipsychotic agent as a mood stabilizer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) score | Baseline, Week 2, Week 8, Week 10, Week 16
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is scored on a scale of 0 to 60, with each of the 10 items rated from 0 to 6 by a trained clinician during an interview. A higher score indicates a more severe level of depression, with common severity ranges being: 0-6 (normal), 7-19 (mild), 20-34 (moderate), and 35-60 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Ozerdem, MD, PhD, Principal Investigator — Mayo Clinic; Deniz Ceylan, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials